CLINICAL TRIAL: NCT00125320
Title: A Phase III Study of the Conversion Efficacy and Safety of Repeated Intravenous Doses of RSD1235 in Subjects With Atrial Fibrillation or Atrial Flutter Following Valvular and/or Coronary Artery Bypass Graft Surgery
Brief Title: Response to RSD1235 Compared to Placebo in Subjects With Atrial Arrhythmia After Heart Surgery
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Collaborators: Astellas Pharma US, Inc. (Industry); Advanz Pharma (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1235-0104
Record Dates: First submitted 2005-07-28; First posted 2005-08-01 (Estimated); Last update posted 2007-12-24 (Estimated); Status verified 2007-12

CONDITIONS: Atrial Fibrillation; Atrial Flutter
Keywords: Treatment
MeSH Terms: conditions — Atrial Fibrillation; Atrial Flutter | interventions — vernakalant

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: RSD1235

SUMMARY:
The purpose of this study is to demonstrate the safety and efficacy of RSD1235 compared to placebo in the conversion of atrial arrhythmia to sinus rhythm in subjects following valvular and/or coronary artery bypass graft surgery.

DETAILED DESCRIPTION:
This multi-national, multi-center study is a double blind, randomized, placebo-controlled trial with 2 parallel treatment arms (1 active, 1 placebo) to assess the conversion efficacy and safety of 2 intravenous doses of RSD1235 in subjects with atrial fibrillation or atrial flutter following valvular and/or coronary artery bypass graft (CABG) surgery.

ELIGIBILITY:
Inclusion Criteria:

* Documented atrial arrhythmia after valvular and/or coronary artery bypass graft surgery

Exclusion Criteria:

* Unstable Class IV heart failure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 190 (Actual)
Dates: Start 2004-06; Primary Completion 2007-02 (Actual); Study Completion 2007-02 (Actual)

PRIMARY OUTCOMES:
Effectiveness of RSD1235 | 90 minutes post infusion

SECONDARY OUTCOMES:
Proportion of patients in sinus rhythm at 90 minutes | Time from first exposure to conversion to sinus rhythm

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Astellas Pharma US, Inc.
Locations (21):
- United States (2):
  - Fort Lauderdale, Florida
  - Atlanta, Georgia
- Argentina (2):
  - Buenos Aires
  - La Plata
- Canada (3):
  - Calgary, Alberta
  - Toronto, Ontario
  - Montreal, Quebec
- Denmark (3):
  - Aalborg, DK
  - Hellerup, DK
  - Odense C, DK
- India (7):
  - Bangalore
  - Chennai
  - Hyderabaad
  - Kerala
  - Mohali
  - Mumbai
  - New Delhi
- Poland (4):
  - Katowice
  - Krakow
  - Lodz
  - Warsaw

REFERENCES:
- [Derived] Kowey PR, Dorian P, Mitchell LB, Pratt CM, Roy D, Schwartz PJ, Sadowski J, Sobczyk D, Bochenek A, Toft E; Atrial Arrhythmia Conversion Trial Investigators. Vernakalant hydrochloride for the rapid conversion of atrial fibrillation after cardiac surgery: a randomized, double-blind, placebo-controlled trial. Circ Arrhythm Electrophysiol. 2009 Dec;2(6):652-9. doi: 10.1161/CIRCEP.109.870204. PMID 19948506